CLINICAL TRIAL: NCT00719186
Title: A 20 Week Double-Blind Randomized Trial of Clomiphene Citrate and Letrozole for the Treatment of Infertility in Women With Polycystic Ovary Syndrome
Brief Title: Pregnancy in Polycystic Ovary Syndrome II
Acronym: PPCOSII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Penn State University (Other); University of Colorado, Denver (Other); University of Michigan (Other); University of Pennsylvania (Other); The University of Texas Health Science Center at San Antonio (Other); University of Vermont (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Heping Zhang, Principal Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RMN-PPCOSII
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-05

CONDITIONS: Pregnancy; Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Infertility; Pregnancy; Women
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Clomiphene; Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Clomiphene citrate 50 mg every day for 5 days (day 3-7 of cycle), for a total of 5 cycles or 20 weeks
  Interventions: Drug: Clomiphene citrate
- B (Active Comparator): Letrozole 2.5 mg every day for 5 days (day 3-7 of cycle), for a total of 5 cycles or 20 weeks
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Clomiphene citrate — Clomiphene citrate 50 mg every day for 5 days (day 3-7 of cycle), for a total of 5 cycles or 20 weeks
  Other Names: Clomid; Serophene
  Arms: A
Drug: Letrozole — Letrozole 2.5 mg every day for 5 days (day 3-7 of cycle), for a total of 5 cycles or 20 weeks
  Other Names: Femara
  Arms: B

SUMMARY:
The primary research hypothesis is that ovulation induction with an aromatase inhibitor (letrozole) is more likely to result in live birth than ovulation induction with a selective estrogen receptor modulator (clomiphene citrate) in infertile women with PCOS. A safety hypothesis will also be incorporated into the primary research hypothesis in which we hypothesize both treatments are equally safe for mother and child.

Secondary research hypotheses include:

1. Treatment with letrozole is more likely to result in singleton pregnancy compared to treatment with clomiphene citrate. Singleton pregnancy is defined as presence of a single intrauterine gestational sac with a single fetal pole and observable heart motion.
2. Treatment with letrozole will less likely result in a first trimester intrauterine fetal demise than treatment with clomiphene citrate. A first trimester IUFD is defined as a pregnancy that ends before 13 weeks gestation.
3. Treatment with letrozole is more likely to result in ovulation (increased ovulation rate) compared to treatment with clomiphene citrate. Ovulation is defined as a midluteal progesterone level ≥ 3 ng/mL.
4. The shortest time to pregnancy will be with letrozole.
5. Age, body mass index, SHBG, testosterone, LH, Anti-Mullerian Hormone (AMH), and degree of hirsutism and acne will be significant predictors of ovulation and conception regardless of treatment.
6. Improvement in SHBG, testosterone, AMH, and LH levels will be significant predictors of ovulation and conception regardless of treatment.
7. DNA polymorphisms in estrogen action genes will predict response to study drug.
8. Quality of Life will be better on letrozole than clomiphene.
9. Letrozole will be more cost effective at achieving singleton pregnancies than clomiphene.

DETAILED DESCRIPTION:
Preliminary data are promising for the use of letrozole to induce ovulation in infertile women with PCOS. However the true magnitude of the effect of letrozole is difficult to discern from prior studies. Therefore we intend to determine the safety and efficacy of letrozole, an aromatase inhibitor, compared to clomiphene citrate, a selective estrogen receptor modulator, in achieving live birth in infertile women with PCOS.

Treatment- After progestin withdrawal, 750 women will be equally randomized to two different treatment arms: A) clomiphene citrate 50 mg every day for 5 days (day 3-7 of cycle), or B) letrozole 2.5 mg every day for 5 days (day 3-7 of cycle), for a total of 5 cycles or 20 weeks. Dose will be increased in subsequent cycles in both treatment groups for non-response or poor ovulatory response up to a maximum of 150 mg of clomiphene a day (x 5 days) or 7.5 mg of letrozole a day (x 5 days).

Statistical Analysis- The primary analysis will use an intent-to-treat approach to examine differences in the live birth rate in the two treatment arms.

Anticipated time to completion- A total of 4 years will be required to complete the study after start up; 31 month enrollment period, 5 month treatment period, with 9 month additional observation to determine pregnancy outcomes. This will be accomplished by enrolling ~3.45 women with PCOS per center per month over the enrollment period (N = 7 RMN sites).

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria (Must have ovulatory dysfunction and either hyperandrogenism or PCO)

1. Chronic anovulation or oligomenorrhea: defined as spontaneous intermenstrual periods of ≥45 days or a total of ≤8 menses per year, or for women with suspected anovulatory bleeding, a midluteal serum progesterone level < 3 ng/mL is indicative of chronic anovulation. For women who have been on ovarian suppressive therapy or other confounding medication (i.e. insulin sensitizing agents) within the last year prior to the study, a history of ≤8 menses per year prior to the initiation of this prior therapy will qualify as evidence of oligomenorrhea. For women with more regular bleeding patterns, but who are suspected to be experiencing anovulatory bleeding, a midluteal progesterone level < 3ng/mL will be evidence of ovulatory dysfunction and qualify as anovulation. Undiagnosed persistent vaginal bleeding should be diagnosed and treated prior to enrollment.
2. Hyperandrogenism (either Hirsutism or Hyperandrogenemia) or Polycystic Ovaries on Ultrasound:

   1. Hirsutism is determined by a modified Ferriman-Gallwey Score >8 at screening exam (Hatch, Rosenfield et al. 1981 Aug 1). Subjects who have hirsutism do not need local or core labs documenting elevated androgen levels.
   2. Hyperandrogenemia can be determined from local labs. Local cutoffs will be pre-determined by each site prior to study initiation. Hyperandrogenemia will be defined as an elevated total testosterone, or free androgen index (FAI)(in our lab at Penn State College of Medicine a total T > 50 ng/dL or a free androgen index >5) will allow entry into the study (Legro, Driscoll et al. 1998). The FAI is calculated from measurable values for total T and SHBG, as previously described (Miller, Rosner et al. 2004), using the following equation: (FAI = Total testosterone in nmol/L / SHBG in nmol/L) X 100. Outside lab values obtained within the last year documenting elevated T or FAI levels are sufficient to meet criteria of hyperandrogenemia.
   3. Polycystic Ovaries on Ultrasound: We will use the revised Rotterdam criteria for diagnosing polycystic ovaries (Balen, Laven et al. 2003). PCO will be defined as either an ovary that contains 12 or more follicles measuring 2-9 mm in diameter, or an increased ovarian volume (> 10 cm3) on one ovary for entry into the study. If there is a follicle > 10 mm in diameter, the scan should be repeated at a time of ovarian quiescence in order to calculate volume and area if the subject does not otherwise qualify for the study. The presence of a single polycystic ovary (PCO), either by volume or morphology, is sufficient to provide the diagnosis.

Exclusion Criteria:

We will exclude subjects with medical conditions that represent contraindications to CC, aromatase inhibitors and/or pregnancy or who are unable to comply with the study procedures. We will exclude subjects with poorly controlled Type I or Type II diabetes; undiagnosed liver disease or dysfunction (based on serum liver enzyme testing); renal disease or abnormal serum renal function; significant anemia; history of deep venous thrombosis, pulmonary embolus, or cerebrovascular accident; uncontrolled hypertension, known symptomatic heart disease; history of or suspected cervical carcinoma, endometrial carcinoma, or breast carcinoma; undiagnosed vaginal bleeding, and use of other medications known to affect reproductive function or metabolism (e.g., OCP, GnRH agonists and antagonists, antiandrogens, gonadotropins, anti-obesity drugs, somatostatin, diazoxide, ACE inhibitors, and calcium channel blockers). As in PPCOS we will allow a 2 months washout period for subjects who desire to participate and discontinue exclusionary medications (most commonly OCP, but also possibly metformin), and a period of observation or treatment for correctable conditions.

Couple Inclusion Criteria

1. Sperm concentration of 14 million/mL in at least one ejaculate within the last year, with at least some motile sperm.
2. Ability to have regular intercourse during the ovulation induction phase of the study.
3. At least one patent tube and normal uterine cavity as determined by sonohysterogram, hysterosalpingogram, or hysteroscopy/laparoscopy within the last 3 years. An uncomplicated intrauterine non-IVF pregnancy and uncomplicated delivery and postpartum course resulting in live birth within the last three years will also serve as sufficient evidence of a patent tube and normal uterine cavity as long as the subject did not have, during the pregnancy or subsequently, risk factors for Asherman's syndrome or tubal disease or other disorder leading to an increased suspicion for intrauterine abnormality or tubal occlusion.
4. No previous sterilization procedures (vasectomy, tubal ligation) that have been reversed. The prior procedure may affect study outcomes.

Specific Exclusion Criteria

1. Current pregnancy.
2. Patients on oral contraceptives, depo-progestins, or hormonal implants (including Implanon). A two month washout period will be required prior to screening for patients on these agents. Longer washouts may be necessary for certain depot contraceptive forms or implants, especially where the implants are still in place. A one-month washout will be required for patients on oral cyclic progestins.
3. Patients with hyperprolactinemia (defined as two prolactin levels at least one week apart > 30 ng/mL or as determined by local normative values). The goal of eliminating patients with documented hyperprolactinemia is to decrease the heterogeneity of the PCOS population. These patients may be candidates for ovulation induction with alternate regimens (dopamine agonists). A normal level within the last year or on treatment is adequate for entry.
4. Patients with known 21-hydroxylase deficiency or other enzyme deficiency leading to the phenotype of congenital adrenal hyperplasia. 21-hydroxylase deficiency will be excluded in all patients by a fasting 17-hydroxyprogesterone (17-OHP) level <2 ng/mL (Azziz, Hincapie et al. 1999 Nov). If relevant, this level should be determined in the follicular phase, because the 17-hydroxyprogesterone level is likely to be elevated beyond this range if the patient is in the luteal phase of an infrequent ovulatory cycle. In the case of elevated fasting 17-OHP levels in the follicular phase, an ACTH stimulation test will be performed. A 1-hour stimulated value > 10 ng/mL will be an exclusion (Moran, Knochenhauer et al. 1998). As 21-hydroxylase deficiency is a congenital condition, any normal level in the past of 17-hydroxyprogesterone allows entry into this study.
5. Patients with menopausal levels of FSH (> 15 mIU/mL). A normal level within the last year is adequate for entry.
6. Patients with uncorrected thyroid disease (defined as TSH < 0.2 mIU/mL or >5.5 mIU/mL). A normal level within the last year is adequate for entry.
7. Patients diagnosed with Type I or Type II diabetes who are poorly controlled (defined as a glycohemoglobin level > 7.0%), or patients receiving antidiabetic medications such as insulin, thiazolidinediones, acarbose, or sulfonylureas likely to confound the effects of study medication; patients currently receiving metformin XR for a diagnosis of Type I or Type II diabetes or for PCOS are also specifically excluded.
8. Patients with liver disease defined as AST or ALT > 2 times normal or total bilirubin >2.5 mg/dL.
9. Patients with renal disease defined as BUN > 30 mg/dL or serum creatinine> 1.4 mg/dL.
10. Patients with significant anemia (Hemoglobin < 10 g/dL).
11. Patients with a history of deep venous thrombosis, pulmonary embolus, or cerebrovascular accident.
12. Patients with known heart disease that is likely to be exacerbated by pregnancy.
13. Patients with a history of, or suspected cervical carcinoma, endometrial carcinoma, or breast carcinoma. A normal Pap smear result within ACOG guidelines for Pap smear frequency will be required for women 21 and over.
14. Patients with a current history of alcohol abuse. Alcohol abuse is defined as > 14 drinks/week or binge drinking.
15. Patients enrolled simultaneously into other investigative studies that require medications, proscribe the study medications, limit intercourse, or otherwise prevent compliance with the protocol. Patients who anticipate taking longer than a one month break during the protocol should not be enrolled.
16. Patients taking other medications known to affect reproductive function or metabolism. These medications include oral contraceptives, GnRH agonists and antagonists, antiandrogens, gonadotropins, anti-obesity drugs, anti-diabetic drugs such as metformin and thiazolidinediones, somatostatin, diazoxide, ACE inhibitors, and calcium channel blockers. The washout period on all these medications will be two months and a list is found in the appendix.
17. Patients with a suspected adrenal or ovarian tumor secreting androgens.
18. Patients with suspected Cushing's syndrome.
19. Couples with previous sterilization procedures (vasectomy, tubal ligation) which have been reversed. The prior procedure may affect study outcomes, and patients with both a reversed sterilization procedure and PCOS are rare enough that exclusion should not adversely affect recruitment.
20. Subjects who have undergone a bariatric surgery procedure in the recent past (<12 months) and are in a period of acute weight loss or have been advised against pregnancy by their bariatric surgeon.
21. Patients with untreated poorly controlled hypertension defined as a systolic blood pressure ≥ 160 mm Hg or a diastolic ≥ 100 mm Hg obtained on two measures obtained at least 60 minutes apart.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 750 (Actual)
Dates: Start 2009-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Eisenberg, MD, MPH, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Nanette Santoro, MD, Study Chair — Albert Einstein College of Medicine; Richard Legro, MD, Principal Investigator — Pennsylvania State University College of Medicine; Robert Brzyski, MD, PhD, Study Director — The University of Texas Health Science Center at San Antonio; Peter Casson, MD, Study Director — University of Vermont; Michael Diamond, MD, Study Director — Wayne State University; Heping Zhang, PhD, Study Director — Yale University; Gregory M Christman, MD, Study Director — University of Michigan; Christos Coutifaris, MD, Study Director — University of Pennsylvania; William D Schlaff, MD, Study Director — University of Colorado Denver Health Science Center
Locations (12):
- United States (12):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Stanford University Medical Center, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Carolinas Medical Center, Charlotte, North Carolina
  - Pennsylvania State University College of Medicine, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Vermont, Burlington, Vermont
  - Virginia Commonwealth University, School of Medicine, Richmond, Virginia

REFERENCES:
- [Derived] Kuokkanen S, Seungdamrong A, Santoro N, Lieman H, Sun F, Wild R, Zhang H, Pal L. A relook at the relevance of thyroid stimulating hormone and thyroid autoimmunity for pregnancy outcomes: Analyses of randomized control trials data from Pregnancy in Polycystic Ovary Syndrome and Assessment of Multiple Intrauterine Gestations from Ovarian Stimulation. Fertil Steril. 2025 May;123(5):873-882. doi: 10.1016/j.fertnstert.2024.12.005. Epub 2024 Dec 12. PMID 39672366
- [Derived] Souter I, Sun F, Zhang H, Diamond MP, Legro RS, Wild RA, Hansen KR, Santoro N; Eunice Kennedy Schriver National Institute of Child Health and Human Development Reproductive Medicine Network. A personalized medicine approach to ovulation induction/ovarian stimulation: development of a predictive model and online calculator from level-I evidence. Fertil Steril. 2022 Feb;117(2):408-418. doi: 10.1016/j.fertnstert.2021.10.024. PMID 35125179
- [Derived] Eisenberg E, Legro RS, Diamond MP, Huang H, O'Brien LM, Smith YR, Coutifaris C, Hansen KR, Santoro N, Zhang H. Sleep Habits of Women With Infertility. J Clin Endocrinol Metab. 2021 Oct 21;106(11):e4414-e4426. doi: 10.1210/clinem/dgab474. PMID 34180998
- [Derived] Engmann L, Sun F, Legro RS, Diamond MP, Zhang H, Santoro N; Reproductive Medicine Network. Factors associated with study protocol adherence and bio banking participation in reproductive medicine clinical trials and their relationship to live birth. Hum Reprod. 2020 Dec 1;35(12):2819-2831. doi: 10.1093/humrep/deaa232. PMID 33190149
- [Derived] Butts SF, Seifer DB, Koelper N, Senapati S, Sammel MD, Hoofnagle AN, Kelly A, Krawetz SA, Santoro N, Zhang H, Diamond MP, Legro RS; Eunice Kennedy Shriver National Institute of Child Health and Human Development Reproductive Medicine Network. Vitamin D Deficiency Is Associated With Poor Ovarian Stimulation Outcome in PCOS but Not Unexplained Infertility. J Clin Endocrinol Metab. 2019 Feb 1;104(2):369-378. doi: 10.1210/jc.2018-00750. PMID 30085176
- [Derived] Greenwood EA, Pasch LA, Cedars MI, Legro RS, Huddleston HG; Eunice Kennedy Shriver National Institute of Child Health and Human Development Reproductive Medicine Network. Association among depression, symptom experience, and quality of life in polycystic ovary syndrome. Am J Obstet Gynecol. 2018 Sep;219(3):279.e1-279.e7. doi: 10.1016/j.ajog.2018.06.017. Epub 2018 Jun 30. PMID 29969586
- [Derived] Evans-Hoeker EA, Eisenberg E, Diamond MP, Legro RS, Alvero R, Coutifaris C, Casson PR, Christman GM, Hansen KR, Zhang H, Santoro N, Steiner AZ; Reproductive Medicine Network. Major depression, antidepressant use, and male and female fertility. Fertil Steril. 2018 May;109(5):879-887. doi: 10.1016/j.fertnstert.2018.01.029. PMID 29778387
- [Derived] Seungdamrong A, Steiner AZ, Gracia CR, Legro RS, Diamond MP, Coutifaris C, Schlaff WD, Casson P, Christman GM, Robinson RD, Huang H, Alvero R, Hansen KR, Jin S, Eisenberg E, Zhang H, Santoro N; Eunice Kennedy Shriver National Institute of Child Health and Human Development Reproductive Medicine Network. Preconceptional antithyroid peroxidase antibodies, but not thyroid-stimulating hormone, are associated with decreased live birth rates in infertile women. Fertil Steril. 2017 Oct 25:S0015-0282(17)31748-X. doi: 10.1016/j.fertnstert.2017.08.026. Online ahead of print. PMID 29102040
- [Derived] Santoro N, Eisenberg E, Trussell JC, Craig LB, Gracia C, Huang H, Alvero R, Casson P, Christman G, Coutifaris C, Diamond M, Jin S, Legro RS, Robinson RD, Schlaff WD, Zhang H; Reproductive Medicine Network Investigators. Fertility-related quality of life from two RCT cohorts with infertility: unexplained infertility and polycystic ovary syndrome. Hum Reprod. 2016 Oct;31(10):2268-79. doi: 10.1093/humrep/dew175. Epub 2016 Jul 7. PMID 27402910
- [Derived] Legro RS, Dodson WC, Kunselman AR, Stetter CM, Kris-Etherton PM, Williams NI, Gnatuk CL, Estes SJ, Allison KC, Sarwer DB, Diamond MP, Schlaff WD, Casson PR, Christman GM, Barnhart KT, Bates GW, Usadi R, Lucidi S, Baker V, Zhang H, Eisenberg E, Coutifaris C, Dokras A. Benefit of Delayed Fertility Therapy With Preconception Weight Loss Over Immediate Therapy in Obese Women With PCOS. J Clin Endocrinol Metab. 2016 Jul;101(7):2658-66. doi: 10.1210/jc.2016-1659. Epub 2016 May 12. PMID 27172435
- [Derived] Steiner AZ, Diamond MP, Legro RS, Schlaff WD, Barnhart KT, Casson PR, Christman GM, Alvero R, Hansen KR, Geisler WM, Thomas T, Santoro N, Zhang H, Eisenberg E; Reproductive Medicine Network. Chlamydia trachomatis immunoglobulin G3 seropositivity is a predictor of reproductive outcomes in infertile women with patent fallopian tubes. Fertil Steril. 2015 Dec;104(6):1522-6. doi: 10.1016/j.fertnstert.2015.08.022. Epub 2015 Sep 25. PMID 26413816
- [Derived] Kuang H, Jin S, Thomas T, Engmann L, Hansen KR, Coutifaris C, Casson P, Christman G, Alvero R, Santoro N, Eisenberg E, Diamond MP, Legro RS, Zhang H; Reproductive Medicine Network. Predictors of participant retention in infertility treatment trials. Fertil Steril. 2015 Nov;104(5):1236-43.e1-2. doi: 10.1016/j.fertnstert.2015.08.001. Epub 2015 Sep 3. PMID 26354094
- [Derived] Kuang H, Jin S, Hansen KR, Diamond MP, Coutifaris C, Casson P, Christman G, Alvero R, Huang H, Bates GW, Usadi R, Lucidi S, Baker V, Santoro N, Eisenberg E, Legro RS, Zhang H; Reproductive Medicine Network. Identification and replication of prediction models for ovulation, pregnancy and live birth in infertile women with polycystic ovary syndrome. Hum Reprod. 2015 Sep;30(9):2222-33. doi: 10.1093/humrep/dev182. Epub 2015 Jul 22. PMID 26202922
- [Derived] Legro RS, Chen G, Kunselman AR, Schlaff WD, Diamond MP, Coutifaris C, Carson SA, Steinkampf MP, Carr BR, McGovern PG, Cataldo NA, Gosman GG, Nestler JE, Myers ER, Zhang H, Foulds J; Reproductive Medicine Network. Smoking in infertile women with polycystic ovary syndrome: baseline validation of self-report and effects on phenotype. Hum Reprod. 2014 Dec;29(12):2680-6. doi: 10.1093/humrep/deu239. Epub 2014 Oct 16. PMID 25324541
- [Derived] Legro RS, Brzyski RG, Diamond MP, Coutifaris C, Schlaff WD, Casson P, Christman GM, Huang H, Yan Q, Alvero R, Haisenleder DJ, Barnhart KT, Bates GW, Usadi R, Lucidi S, Baker V, Trussell JC, Krawetz SA, Snyder P, Ohl D, Santoro N, Eisenberg E, Zhang H; NICHD Reproductive Medicine Network. Letrozole versus clomiphene for infertility in the polycystic ovary syndrome. N Engl J Med. 2014 Jul 10;371(2):119-29. doi: 10.1056/NEJMoa1313517. PMID 25006718
- [Derived] Legro RS, Brzyski RG, Diamond MP, Coutifaris C, Schlaff WD, Alvero R, Casson P, Christman GM, Huang H, Yan Q, Haisenleder DJ, Barnhart KT, Bates GW, Usadi R, Lucidi R, Baker V, Trussell JC, Krawetz SA, Snyder P, Ohl D, Santoro N, Eisenberg E, Zhang H; National Institute of Child Health and Human Development Reproductive Medicine Network. The Pregnancy in Polycystic Ovary Syndrome II study: baseline characteristics and effects of obesity from a multicenter randomized clinical trial. Fertil Steril. 2014 Jan;101(1):258-269.e8. doi: 10.1016/j.fertnstert.2013.08.056. Epub 2013 Oct 21. PMID 24156957
- [Derived] Schlaff WD, Zhang H, Diamond MP, Coutifaris C, Casson PR, Brzyski RG, Christman GM, Barnhart KT, Trussell JC, Krawetz SA, Snyder PJ, Ohl D, Santoro N, Eisenberg E, Huang H, Legro RS; Reproductive Medicine Network. Increasing burden of institutional review in multicenter clinical trials of infertility: the Reproductive Medicine Network experience with the Pregnancy in Polycystic Ovary Syndrome (PPCOS) I and II studies. Fertil Steril. 2011 Jul;96(1):15-8. doi: 10.1016/j.fertnstert.2011.05.069. Epub 2011 Jun 8. PMID 21645894
- See also: Related Info — http://c2s2.yale.edu/rmn/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Clomiphene Citrate: Clomiphene citrate 50 mg every day for 5 days (day 3-7 of cycle), for a total of 5 cycles or 20 weeks
  Clomiphene citrate: Clomiphene citrate 50 mg every day for 5 days (day 3-7 of cycle), for a total of 5 cycles or 20 weeks
- Arm B: Letrozole: Letrozole 2.5 mg every day for 5 days (day 3-7 of cycle), for a total of 5 cycles or 20 weeks
  Letrozole: Letrozole 2.5 mg every day for 5 days (day 3-7 of cycle), for a total of 5 cycles or 20 weeks
Period: Overall Study
Arm/Group | Arm A: Clomiphene Citrate | Arm B: Letrozole
Started | 376 | 374
Completed | 376 | 374
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Clomiphene Citrate | Arm B: Letrozole | Total
Number analyzed (Participants) | 376 | 374 | 750
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (4.0) | 28.9 (4.5) | 28.9 (4.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 376 | 374 | 750
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 376 | 374 | 750
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 376 | 374 | 750

OUTCOME MEASURES:

1. Primary Outcome: Live Birth
Description: The primary outcome measure is the occurrence of a live birth during the study period. Safety measures will be the number and type of reported adverse events in subjects and offspring.
Time Frame: as few as 5 months, up to 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Clomiphene Citrate | Arm B: Letrozole
Number analyzed (Participants) | 376 | 374
Participants | 72 | 103
Statistical Analysis 1: Comparison: Arm A: Clomiphene Citrate vs Arm B: Letrozole; Test type: Superiority or Other; p = 0.007, Chi-squared

2. Secondary Outcome: Number of Pregnancy
Time Frame: as few as 5 months, up to 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Clomiphene Citrate | Arm B: Letrozole
Number analyzed (Participants) | 376 | 374
Participants | 103 | 154

3. Secondary Outcome: Number of Ovulations
Time Frame: as few as 5 months, up to 16 months
Measure: Number; unit: ovulations
Arm/Group | Arm A: Clomiphene Citrate | Arm B: Letrozole
Number analyzed (Participants) | 376 | 374
ovulations | 331 | 388

4. Secondary Outcome: Number of Serious Adverse Events
Time Frame: as few as 5 months, up to 16 months
Measure: Number; unit: events
Arm/Group | Arm A: Clomiphene Citrate | Arm B: Letrozole
Number analyzed (Participants) | 376 | 374
events | 13 | 22

5. Secondary Outcome: Neonatal Complication Rate
Time Frame: September 2008 - December 2011
Population: Neonatal complications reported per infant, an infant could have more than one complication.
Measure: Number; unit: participants
Arm/Group | Arm A: Clomiphene Citrate | Arm B: Letrozole
Number analyzed (Participants) | 66 | 102
participants
  Neonatal jaundice | 17 | 27
  Neonatal respiratory distress syndrome | 2 | 7
  Neonatal hospitalization >3 days | 4 | 4
  Intrauterine growth restriction | 1 | 5
  Neonatal infectin | 2 | 2
  Minor birth defect | 0 | 1
  Other complication | 4 | 5
  Congenital anomaly | 1 | 4
  Neonatal death | 2 | 1

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Arm A: Clomiphene Citrate | Arm B: Letrozole
Serious Adverse Events (participants affected / at risk) | 13/376 | 21/374
Other Adverse Events (participants affected / at risk) | 283/355 | 285/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Clomiphene Citrate (N=376) | Arm B: Letrozole (N=374)
Ovarian torsion (Reproductive system and breast disorders) | 1 | 0
Ectopic Pregnancy (Reproductive system and breast disorders) | 3 | 4
Ruptured Corpus Luteum Cyst (Reproductive system and breast disorders) | 0 | 1
Carcinoma of the Skin-stage 3 (Skin and subcutaneous tissue disorders) | 1 | 0
cholecystectomy (Hepatobiliary disorders) | 1 | 1
Heterotopic Pregnancy (Reproductive system and breast disorders) | 1 | 0
Pregnancy of Unknown Location (Reproductive system and breast disorders) | 1 | 1
Appendectomy (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Mid ureteral stone (Renal and urinary disorders) | 0 | 1
Congenital Anomaly (Congenital, familial and genetic disorders) | 1 | 4
Fetal Demise (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Neonatal death (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Hospitalization (General disorders) | 3 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Clomiphene Citrate (N=355) | Arm B: Letrozole (N=359)
Headache (Nervous system disorders) | 170 | 167
abdominal/pelvic pain (Musculoskeletal and connective tissue disorders) | 138 | 146
Nausea (Gastrointestinal disorders) | 91 | 110
Hot flashes (Endocrine disorders) | 117 | 73
Breast pain (Reproductive system and breast disorders) | 76 | 76
Fatigue (General disorders) | 53 | 78
Dysmenorrhea (Reproductive system and breast disorders) | 64 | 60
Back pain (Musculoskeletal and connective tissue disorders) | 55 | 64
Dyspepsia (Gastrointestinal disorders) | 62 | 45
Abdominal bloating (Gastrointestinal disorders) | 42 | 49
Agitation (Psychiatric disorders) | 37 | 43
Dizziness (Nervous system disorders) | 27 | 44
Upper respiratory infection (Infections and infestations) | 31 | 38
Irritability (Psychiatric disorders) | 33 | 33
Joint/limb pain (Musculoskeletal and connective tissue disorders) | 26 | 33
Flu like symptoms (Infections and infestations) | 18 | 29
Diarrhea (Gastrointestinal disorders) | 18 | 24
Vomiting (Gastrointestinal disorders) | 20 | 21
Acne/ oily skin (Skin and subcutaneous tissue disorders) | 24 | 16
Constipation (Gastrointestinal disorders) | 20 | 17
Abnormal vaginal bleeding (Reproductive system and breast disorders) | 9 | 18
Insomnia (Psychiatric disorders) | 14 | 12
Vaginal infection (Infections and infestations) | 16 | 8
Allergic rhinitis (Infections and infestations) | 12 | 10
fever (Infections and infestations) | 9 | 13
Urinary tract infection (Infections and infestations) | 10 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 10
Depression (Psychiatric disorders) | 10 | 6
Urinary frequency (Renal and urinary disorders) | 8 | 7
Vaginal discharge (Reproductive system and breast disorders) | 4 | 9
Blurred vision (Eye disorders) | 4 | 8
Chills (General disorders) | 8 | 4
Sinus complaints (Respiratory, thoracic and mediastinal disorders) | 4 | 8
First Trimester other complication during pregnancy (General disorders) | 8 | 15
Second Trimester Hyperemesis (Pregnancy, puerperium and perinatal conditions) | 5 | 8
Second Trimester Gestational Diabetes (Pregnancy, puerperium and perinatal conditions) | 13 | 27
Second Trimester Pre-eclampsia/ eclampsia (Pregnancy, puerperium and perinatal conditions) | 13 | 18
Second Trimester pretem labor (Pregnancy, puerperium and perinatal conditions) | 12 | 14
Second Trimester Premature rupture of membrane (Pregnancy, puerperium and perinatal conditions) | 7 | 8
Second Trimester Incompetant cervix (Pregnancy, puerperium and perinatal conditions) | 6 | 8
Post-partum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 3 | 8
Post-partum Infection (Infections and infestations) | 2 | 7
Neonatal Jaundice (Hepatobiliary disorders) | 17 | 27
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No